CLINICAL TRIAL: NCT05277766
Title: Intraperitoneal Aerosolized Nanoliposomal Irinotecan (Nal-IRI) in Peritoneal Carcinomatosis From Gastrointestinal Cancer: a Phase I Study
Brief Title: Intraperitoneal Aerosolized Nanoliposomal Irinotecan (Nal-IRI) in Peritoneal Carcinomatosis From Gastrointestinal Cancer
Acronym: PIPAC-NAL-IRI
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Kom Op Tegen Kanker (Other); University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ONZ-2022-0120
Record Dates: First submitted 2022-02-18; First posted 2022-03-14 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Peritoneal Carcinomatosis; Peritoneal Metastases; Colorectal Cancer; Small Bowel Cancer; Appendix Cancer; Gastric Cancer; Pancreatic Cancer; Bile Duct Cancer
Keywords: PIPAC; Nal-IRI; Peritoneal carcinomatosis; dose-finding study; pharmacokinetics; pharmacodynamics; safety and efficacy; Onivyde; Primary gastrointestinal cancer; Colorectal cancer; Small bowel cancer; Appendix cancer; Stomach cancer; Pancreatic cancer; Cholangiocarcinoma; dose-escalation study; Peritoneal metastases
MeSH Terms: conditions — Peritoneal Neoplasms; Colorectal Neoplasms; Appendiceal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Bile Duct Neoplasms; Cholangiocarcinoma | interventions — irinotecan sucrosofate

STUDY DESIGN:
Intervention Model Description: Phase I study with dose escalation according to two-stage time-to-event continual reassessment method (TITE-CRM): 3x30 - 3x45 - 4x60 - 4x 75 - 16x90 mg/m2 (number of patients x assigned dose). Dose escalation is continued until dose-limiting toxicity (DLT) is observed. Only DLTs that take place within 14 weeks of the start of the treatment are considered.
  From that moment, TITE-CRM updates an initial prior estimate of the probabilities of DLT based on all available information, including patients with incomplete follow-up. Newly accrued patients are assigned the dose whose estimated probability of DLT at that time is closest to target probability. This method allows for continuous, staggered accrual of patients. The target-probability of DLT is 30%. The estimated MTD will be the dose whose estimated posterior probability of DLT is closest to that targeted probability.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Nal-IRI (Onivyde) - 30mg/m² (Experimental): PIPAC with Onivyde (30 mg/m²) will be administered every 4 to 6 weeks for 3 cycles.
  Interventions: Drug: PIPAC with Nal-IRI
- Nal-IRI (Onivyde) - 45mg/m² (Experimental): PIPAC with Onivyde (45 mg/m²) will be administered every 4 to 6 weeks for 3 cycles.
  Interventions: Drug: PIPAC with Nal-IRI
- Nal-IRI (Onivyde) - 60mg/m² (Experimental): PIPAC with Onivyde (60 mg/m²) will be administered every 4 to 6 weeks for 3 cycles.
  Interventions: Drug: PIPAC with Nal-IRI
- Nal-IRI (Onivyde) - 75mg/m² (Experimental): PIPAC with Onivyde (75 mg/m²) will be administered every 4 to 6 weeks for 3 cycles.
  Interventions: Drug: PIPAC with Nal-IRI
- Nal-IRI (Onivyde) - 90mg/m² (Experimental): PIPAC with Onivyde (90 mg/m²) will be administered every 4 to 6 weeks for 3 cycles.
  Interventions: Drug: PIPAC with Nal-IRI

INTERVENTIONS:
Drug: PIPAC with Nal-IRI — Nanoliposomal irinotecan (Nal-IRI, Onivyde) will be administered intraperitoneally using the PIPAC technique. The administered dose will escalate ranging from 30 to 90 mg/m². PIPAC will be performed every 4 to 6 weeks for 3 cycles.
  Other Names: Onivyde

SUMMARY:
The PIPAC NAL-IRI study is designed to examine the maximal tolerated dose of nanoliposomal irinotecan (Nal-IRI, Onivyde) administered with repeated pressurized intraperitoneal aerosol chemotherapy (PIPAC), in a monocentric, phase I trial.

DETAILED DESCRIPTION:
Peritoneal metastases (PM) are a common manifestation of gastrointestinal cancer. The prognosis of patients with PM is particularly poor, and response to systemic chemotherapy is worse compared to parenchymal metastatic cancer in the liver or lungs. In addition, patients with PM frequently develop debilitating symptoms such as intractable ascites, bowel obstruction, or ureteric obstruction, resulting in a severely compromised quality of life.

In selected patients with widespread PM, pressurized intraperitoneal aerosol chemotherapy (PIPAC) holds considerable promise. Briefly, PIPAC combines laparoscopy with intraperitoneal (IP) administration of chemotherapy as an aerosol, which is generated by a nebulizer. The pharmacokinetic (PK) and clinical advantages of PIPAC may be further enhanced by using nanosized anticancer drugs. Nal-IRI (Onivyde) is a nanoliposomal formulation of irinotecan (Camptothecin-11 (CPT-11)), with a markedly superior efficacy when compared with free CPT-11 in human breast and colon cancer xenograft models.

This is a phase I clinical study with aerosolized IP Nal-IRI in patients with PM from GI cancer. In this phase I study, dose escalation will be combined with pharmacokinetic/pharmacodynamic modelling which incorporates, in addition to plasma, tumour tissue, and peritoneal drug concentrations, biomarkers of toxicity and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven cancer of the pancreas, gallbladder or biliary tract, stomach, small bowel, colon, rectum, or appendix with extensive or irresectable peritoneal carcinomatosis
* Estimated life expectancy > 6 months; > 3 months if primary cancer is pancreatic
* Age ≥ 18 years
* Adequate performance status (Karnofsky index > 60% and WHO performance status < 2)
* Written informed consent obtained prior any act of the research

Exclusion Criteria:

* Concomitant systemic (IV) treatment with irinotecan (either as monotherapy or as part of a combination regimen such as FOLFIRI, CAPIRI, or FOLFOXIRI)
* Pregnancy or breastfeeding during the clinical study
* Patients of childbearing age unable or unwilling to provide effective contraception during the study and until the end of relevant exposure (extended by 30 days (female participants) or 120 days (male participants) since the IMP is genotoxic).
* Known allergy or intolerance to irinotecan
* Significant amount of ascites detectable (exceeding 3l in volume)
* Intestinal or urinary tract obstruction
* Extensive hepatic and/or extra-abdominal metastatic disease
* Impaired renal function (serum creatinine > 1.5 mg/dl or calculated GFR (CKD-EPI) < 60 mL/min/1.73 m²
* Impaired liver function (serum total bilirubin > 1.5 mg/dl, except for known Gilbert's disease)
* Platelet count < 100.000/µl
* Hemoglobin < 9g/dl
* Neutrophil granulocytes < 1.500/ml
* Patients known to use:

  * CYP3A4 inducers (rifampin, phenytoin, carbamazepine, rifabutin, rifapentine, phenobarbital, St John's wort)
  * inhibitors of CYP3A4 (clarithromycin, indinavir, itraconazole, lopinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telaprevir, voriconazole) or UGT1A1 (atazanavir, gemfibrozil, indinavir, regorafenib)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Maximally tolerated dose (MTD) of Nal-IRI | Within 14 weeks of the start of the treatment
  Dose limiting toxicities will be monitored.

SECONDARY OUTCOMES:
Recommended phase 2 dose | 6 months after last subject's third PIPAC
  Define the dose recommended to use in a follow-up phase 2 trial based on incidence of DLT and toxicity data scored with CTCAE v5.0 for chemotherapy related toxicity.
Surgical morbidity will be measured | 6 months after third PIPAC
  This will be estimated with the Dindo-Clavien classification and the comprehensive complication index (CCI).
Maximum concentration (Cmax) of nanoliposomal irinotecan | Plasma at 10 timepoints: T= pre-dose (0 minutes=start nebulization), T=30 minutes, T=1.5 hour, T=2.5 hours, T=6 hours, T=24 hours, T=72 hours, T=168 hours, T=336 hours, T=504 hours // Tissue: T= pre-dose (0 minutes=start nebulization), T = 30 minutes
  Determined for CPT-11, SN-38 and SN-38G in plasma and tumor tissue using UPLC-MS/MS.
Time to reach maximum concentration (Tmax) of nanoliposomal irinotecan | Plasma at 10 timepoints: T= pre-dose (0 minutes=start nebulization), T=30 minutes, T=1.5 hour, T=2.5 hours, T=6 hours, T=24 hours, T=72 hours, T=168 hours, T=336 hours, T=504 hours // Tissue: T= pre-dose (0 minutes=start nebulization), T = 30 minutes
  Determined for CPT-11, SN-38 and SN-38G in plasma and tumor tissue using UPLC-MS/MS.
Area under the curve (AUC0h-24h) of nanoliposomal irinotecan | Plasma at 10 timepoints: T= pre-dose (0 minutes=start nebulization), T=30 minutes, T=1.5 hour, T=2.5 hours, T=6 hours, T=24 hours, T=72 hours, T=168 hours, T=336 hours, T=504 hours // Tissue: T= pre-dose (0 minutes=start nebulization), T = 30 minutes
  Determined for CPT-11, SN-38 and SN-38G in plasma and tumor tissue using UPLC-MS/MS.
Volume of distribution (Vd) of nanoliposomal irinotecan | Plasma at 10 timepoints: T= pre-dose (0 minutes=start nebulization), T=30 minutes, T=1.5 hour, T=2.5 hours, T=6 hours, T=24 hours, T=72 hours, T=168 hours, T=336 hours, T=504 hours // Tissue: T= pre-dose (0 minutes=start nebulization), T = 30 minutes
  Determined for CPT-11, SN-38 and SN-38G in plasma and tumor tissue using UPLC-MS/MS.
Clearance (Cl) of nanoliposomal irinotecan | Plasma at 10 timepoints: T= pre-dose (0 minutes=start nebulization), T=30 minutes, T=1.5 hour, T=2.5 hours, T=6 hours, T=24 hours, T=72 hours, T=168 hours, T=336 hours, T=504 hours // Tissue: T= pre-dose (0 minutes=start nebulization), T = 30 minutes
  Determined for CPT-11, SN-38 and SN-38G in plasma and tumor tissue using UPLC-MS/MS.
Elimination half-life (T1/2) of nanoliposomal irinotecan | Plasma at 10 timepoints: T= pre-dose (0 minutes=start nebulization), T=30 minutes, T=1.5 hour, T=2.5 hours, T=6 hours, T=24 hours, T=72 hours, T=168 hours, T=336 hours, T=504 hours // Tissue: T= pre-dose (0 minutes=start nebulization), T = 30 minutes
  Determined for CPT-11, SN-38 and SN-38G in plasma and tumor tissue using UPLC-MS/MS.
Pharmacodynamics (PD) of nanoliposomal irinotecan will be analysed with the Peritoneal regression grading score (PRGS) | T= pre-dose (0 minutes= start nebulization)
  Evaluated on tumor biopsies to determine histological treatment response
Pharmacodynamics (PD) of nanoliposomal irinotecan will be analysed by tumor biopsies. | T= 30 minutes
  Tumour samples will be collected at the end of the aerosol delivery after each PIPAC procedure.
Time-to-event endpoints | 12 months after last subjects last visit
  To evaluate patient's follow-up, several time-to-event endpoints are recorded which include: overall survival (OS), progression free survival (PFS) and peritoneal progression free survival (PPFS).
Quality of Life (The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire, EORTC QLQ-C30) | Pre-operatively (every PIPAC), week 2 (every PIPAC) and, at 3 months, 6months and 12 months after last PIPAC procedure
  This will be investigated using the EORTC QLQ-C30 questionnaire. As to question 1 to 28: the scale varies from 1 (not at all) to 4 (very much). A higher value indicates a lower quality of life. The total score will be between 28 and 112.
  The scale of question 29 and 30 varies from 1 (very poor) to 7 (excellent). The higher the value, the better the quality of life. The total score will be between 2 and 14
Quality of Life (Functional Assessment of Cancer Therapy, FACT-G questionnaire) | Pre-operatively (every PIPAC), week 2 (every PIPAC) and, and at 3 months, 6months and 12 months after last PIPAC procedure
  This will be investigated using the FACT-G questionnaire. The scale of all questions varies from 0 (not at all) to 4 (very much). The total score will be between 0 and 108. The lower the total score, the better the quality of life.
Quality of Life (Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE™) score) | Determined before each PIPAC, every 14th day after PIPAC and at 3 months, 6months and 12 months after last PIPAC procedure
  This will be investigated using the PRO-CTCAE™ questionnaire. The scale of all questions varies from 0 to 4 or 0 to 1 representing absent/present. PRO-CTCAE scores for each attribute (frequency, severity and/or interference) should be presented descriptively (eg. summary statistics or graphical presentations).
Pain assessment performed by patient (Visual Analog Scale (VAS), Pain ) | Determined before each PIPAC procedure, one day postoperatively, and one week after the procedure.
  With this score, pain is assessed on a horizontal line, 100 mm in length, anchored by word descriptors at each end, no pain and very severe pain respectively. The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left-hand end of the line to the point that the patient marks.
Overall treatment response | Determined 8 months after last subject last visit
  Determined according to the RECIST criteria, if possible (measurable lesions on CT or MRI). When no target lesions available, overall treatment response (stable disease, partial response, or progressive disease) will be determined by incorporating PRGS, clinical signs and symptoms, tumor markers, imaging findings (other than target lesions, e.g. ascites volume).

OTHER OUTCOMES:
Exploratory outcome: DNA topoisomerase I (TOP-1) gene copy number | 8 months after last subject last visit
  This will be determined in plasma and tissue samples. This outcome evaluates anti-cancer efficacy.
Exploratory outcome: Expression of human carboxylesterase 2 (hCE2) | 8 months after last subject last visit
  This will be determined in plasma and tissue samples. This outcome evaluates conversion of CPT-11 to SN-38 between patients.

CONTACTS AND LOCATIONS:
Overall Officials: Wim P Ceelen, MD, PhD, Prof, Principal Investigator — University Hospital, Ghent
Locations (1):
- UZ Ghent, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No